CLINICAL TRIAL: NCT03448744
Title: A Multicenter, Randomized, Open-label Control Study to Evaluate Efficacy and Safety of Combination Therapy of Thymalfasin and Entecavir in HBeAg-positive ETV-experienced Patients
Brief Title: Efficacy and Safety of Combination Therapy of Thymalfasin and Entecavir in HBeAg-positive ETV-experienced Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wen-hong Zhang (Other)
Responsible Party: Sponsor-Investigator, Wen-hong Zhang, Professor, Huashan Hospital
Organization: Huashan Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KY2016-219
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Chronic Hepatitis b
Keywords: thymosin alpha; entecavir
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — Thymalfasin; entecavir

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- combiantion therapy group (Experimental): thymosin alpha 1 (1.6 mg subcutaneously injection twice a week) plus ETV (0.5 mg orally, daily) for 24 weeks, and followed by continuous ETV for at least 48 weeks
  Interventions: Drug: Thymosin Alpha1; Drug: Entecavir
- entecavir group (Placebo Comparator): ETV (0.5 mg orally, daily) at least for 72 weeks
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Thymosin Alpha1 — Thymosin Alpha1 (1.6 mg subcutaneously injection twice a week) plus ETV (0.5 mg orally, daily) for 24 weeks, and followed by continuous ETV for at least 48 weeks
  Arms: combiantion therapy group
Drug: Entecavir — ETV (0.5 mg orally, daily) for 72 weeks

SUMMARY:
This is a multicenter, randomized, open-label control trial of two arms conducted at 10 centres in China.The aim was to investigate whether sequential combination therapy with Thymosin alpha 1 and entecavir is superior to continuous ETV monotherapy in HBeAg-positive chronic hepatitis B patients with previous long-term entecavir therapy (≥ 2 years), and to select the optimal patients who may benefit from sequential combination therapy.

DETAILED DESCRIPTION:
To investigate whether sequential combination therapy with Thymosin alpha 1 and entecavir is superior to continuous ETV monotherapy in HBeAg-positive chronic hepatitis B patients with previous long-term entecavir therapy (≥ 1 years), and to select the optimal patients who may benefit from sequential combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* HBsAg positive and anti-HBs negative for more than 6 months
* Being currently treated with ETV ≥1 years
* HBeAg positivity and HBV DNA <60IU/mL with HBsAg <1500IU/mL and HBeAg <200S/CO at screening
* ALT ≤5*ULN and total bilirubin ≤2*ULN
* Age ≥ 18 yrs but ≤ 55 yrs
* Written informed consent

Exclusion Criteria:

* Patients who have contraindications for Thymosin alpha 1 in accordance with the approved summary of product characteristics
* Patients with ALT > 5 x ULN or total bilirubin >2*ULN
* Patients with evidence of hepatocellular carcinoma at screening
* Patients with Child-Pugh score ≥7 or had a history of hepatic encephalopathy or esophageal pile or ascites
* Patients with serological evidence of co-infection with hepatitis A virus, hepatitis C, human immunodeficiency virus or hepatitis D virus
* Patients with a history of excessive drinking: male >40g/d,female >40g/d
* Pregnant or breast-feeding women
* A history of liver transplantation or planned for liver transplantation
* Patients of autoimmune disease
* Patients with other diseases combined
* Patients with creatinine >1.5*ULN
* Investigator considered not proper for participating the trial
* Patients with other maliginant tumor

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 240 (Estimated)
Dates: Start 2017-10-25 (Actual); Primary Completion 2018-12-30 (Estimated); Study Completion 2018-12-30 (Estimated)

PRIMARY OUTCOMES:
HBeAg seroconversion rate at week 72 | week 72
  HBeAg seroconversion rate at week 72

SECONDARY OUTCOMES:
HBeAg seroconversion rate at week 48 | week 48
  HBeAg seroconversion rate at week 48
HBsAg loss at week 48 | week 48
  HBsAg loss at week 48
HBsAg loss at week 72 | week 72
  HBsAg loss at week 72
HBsAg seroconversion at week 72 | week 72
  HBsAg seroconversion at week 72
HBsAg seroconversion at week 48 | week 48
  HBsAg seroconversion at week 48
HBsAg decline during the clinical trial | week 12, weeek 24, week 36, week 48 and week 72
  HBsAg decline during the clinical trial
ALT normalization rate at week 72 | week 72
  ALT normalization rate at week 72
ALT normalization rate at week 48 | week 48
  ALT normalization rate at week 48
Rate of HBV DNA <20IU/mL at week 72 | week 72
  Rate of HBV DNA <20IU/mL at week 72
Rate of HBV DNA <20IU/mL at week 48 | week 48
  Rate of HBV DNA <20IU/mL at week 48

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, Ph.D, Principal Investigator — Department of Infectious Diseases, Huashan Hospital
Locations (1):
- Huashan Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No